CLINICAL TRIAL: NCT04496271
Title: Quality Control of CE-Certified Phonak Hearing Aids - 2020_06
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sonova AG (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Other
Other Study IDs: Sonova2020_06
Record Dates: First submitted 2020-02-28; First posted 2020-08-03 (Actual); Last update posted 2022-11-28 (Actual); Status verified 2020-04

CONDITIONS: Hearing Loss
MeSH Terms: conditions — Hearing Loss

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Successor of Phonak Audéo M-90 (Experimental): Phonak Hearing aid with modified precalculation.
  Interventions: Device: RIC (Receiver in channel)- device
- Phonak Audéo M-90 (Active Comparator): Phonak Audéo M-90 is the most recent Receiver In Canal hearing aid by Phonak which will be fitted to the participants individual hearing loss.
  Interventions: Device: RIC (Receiver in channel)- device

INTERVENTIONS:
Device: RIC (Receiver in channel)- device — HI is developed to support hearing impaired people in calm and complex situations and to be able to participate in communication

SUMMARY:
Phonak Hearing Devices pass through different development and study phases. At an early stage, feasibility studies are conducted to investigate new algorithms, features and functions in an isolated manner. If the benefit is proven, their performance is then investigated regarding interdependency between all available algorithms, features and functions running in parallel in a hearing aid (pivotal/pre-validation studies) and, resulting from the pre-validation studies, they get optimized. Prior to product launch, the Phonak Hearing Systems get reviewed by a final quality control in terms of clinical trials. This is a validation study, investigating improved algorithms, features, functions and wearing comfort. This will be a clinical investigation which will be conducted mono centric at Sonova AG Headquarters based in Stäfa (Switzerland).

DETAILED DESCRIPTION:
This study will investigate the combination of the features to determine if the audiological performance and quality of the new successor of the Marvel family shows an improved benefit over Phonak Audéo Marvel before going into the System Validation. Therefore this study will be a comparative study. The study will determine if hearing impaired users wearing the successor hearing aids, have better initial acceptance with the new precalculation, better sound quality and speech intelligibility, more clarity and loudness comfort in soft and loud environments compared to Phonak Marvel RIC (Receiver in channel) hearing aids. Another objective of the study is to compare the listening effort with the two different study devices.

ELIGIBILITY:
Inclusion Criteria:

* Self-reported confidence to using Bluetooth smartphone
* Hearing Loss range: moderate and moderate/ severe
* experienced hearing aid user
* willingness and interest in testing new features
* willingness to wear behind the ear hearing aids
* Informed Consent as documented by signature

Exclusion Criteria:

* the audiogram is not in the fitting range of the intended hearing aid
* limited mobility and not in the position to attend weekly appointments in Stäfa (Switzerland)
* participant is not able to describe experiences and hearing impressions
* participant has finger movement disorders

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2020-01-13 (Actual); Primary Completion 2020-03-16 (Actual); Study Completion 2020-04-08 (Actual)

PRIMARY OUTCOMES:
Rating of the sound quality for the new and the comparative Hearing aid | 5 weeks
  Subjective rating of the overall satisfaction for sound quality by questionnaires for the new HI and the old comparative HI (%). The questionnaire includes rating scales for the satisfaction. The participant has to rate it in percentage (100% = very satisfy, 0% = very unsatisfy)

SECONDARY OUTCOMES:
Rating sound quality of own voice | 5 weeks
  Evaluating subjectively the HI regarding to the naturalness of the own voice. Participant will be ask in the first visit for spontaneous acceptance, regarding to the quality of their own voice, by rating scales. They have to rate the clarity, dullness etc. of their own voice. Also they will be ask after the hometrial how satisfy they are with the sound quality of their own voice.They have to rate it by rating scales in percentage. (e.g. very satisfy = 100%, very unsatisfy = 0%)
Evaluating listening effort | 5 weeks
  Evaluating listening effort by a special feature. The participants will be in a noisy test situation and have to listen to words, which they should repeat. After each group of words they will be ask to rate how difficult it was to understand by a rating scala (very difficult-difficult-somewhat-easy-very easy). The participants have to do that with the new and the old RIC device. The test will be randomized and single blinded.

CONTACTS AND LOCATIONS:
Locations (1):
- Sonova AG, Stäfa, Switzerland

IPD SHARING:
Plan to Share IPD: No